CLINICAL TRIAL: NCT06410677
Title: Prediction of Immune Infiltration Level and Immunotherapy Efficacy of Esophageal Squamous Cell Carcinoma Based on Multimodal Deep Learning
Brief Title: Changhai Multimodal Esophageal Cancer Cohort
Acronym: CMECC
Status: Active, not recruiting | Type: Observational
Sponsor: Wangluowei (Other)
Responsible Party: Sponsor-Investigator, Wangluowei, M.D., PhD., Doctoral supervisor, Professor, Chief physician, Changhai Hospital
Organization: Changhai Hospital (Other)
Other Study IDs: CMECC
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: deep learning; Esophageal Squamous Cell Carcinoma; immune infiltration
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 110 cases of esophageal squamous cell carcinoma patients. The data types include:
  ① H&E stained images: These atlases display the morphology and tissue structure of cells through the staining of tissue sections, providing important morphological information for disease research.
  ② Molecular data: Molecular information obtained using NanoString technology reveals changes in gene expression, providing a data foundation for the study of the molecular mechanisms of the disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- esophageal squamous cell carcinoma
  Interventions: Diagnostic Test: DNA Sequencing, RNA Sequencing

INTERVENTIONS:
Diagnostic Test: DNA Sequencing, RNA Sequencing — High-coverage Whole-Exome Sequencing sequencing of DNA samples from ESCC was performed.
  RNA expression was analyzed using the NanoString PanCancer Immuno-Oncology 360TM Panel that includes a set of more than 700 genes involved in the main biological pathways of human immunity. These experiments were performed by the Genomics platform of Institut Curie. Total RNAs were used as templates.

SUMMARY:
The burden of esophageal squamous cell carcinoma (ESCC) in China is substantial, with 85% of the cancers being in the progressive stage. The treatment for advanced ESCC are extremely limited, and immunotherapy, represented by PD-1 inhibitors, has demonstrated a promising application potential. However, the effectiveness of PD-1 inhibitors varies significantly among patients with different types of ESCC, and currently, there is no effective method to predict the response to PD-1 inhibitors. In this study, investigators aim to construct a multimodal deep learning-based model to predict the level of immune infiltration and the efficacy of immunotherapy for ESCC, integrating both pathological image features and clinical information of patients with ESCC, thereby enhancing the level of individualized and precise treatment for ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of Hematoxylin and Eosin (H&E) stained images, molecular data obtained through RNA sequencing (RNA-Seq, DNA-seq), and comprehensive clinical information including patient age, gender, history of alcohol consumption, history of smoking, AJCC Tumor, Node, Metastasis Stage, specific location of oesophageal cancer occurrence, and history of reflux.
2. The sample collection is restricted to cancerous tissue, encompassing both primary tumor samples and those from metastatic sites.

Exclusion Criteria:

1. Patients diagnosed with adenosquamous carcinoma or presenting with a combination of other types of oesophageal cancers;
2. Cases involving combined adenocarcinoma affecting the gastroesophageal junction;
3. Individuals with high-grade tumors that have not penetrated the basement membrane, as confirmed by postoperative pathological examination;
4. Subjects in whom postoperative pathology confirms an absence of residual malignant tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 110 patients with ESCC in the Changhai hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Immunogene signatures with predictive value for immunotherapy of ESCC | After undergoes surgery.

SECONDARY OUTCOMES:
Prognosis and immunotherapy tolerance in ESCC patients | Follow-up for at least 1 year after undergoing surgery
  The prognosis was determined through follow-up, while tolerance to immunotherapy was anticipated utilizing gene sequencing methodologies.

CONTACTS AND LOCATIONS:
Overall Officials: Luowei Wang, Study Chair — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
A planned initiative that includes sharing DNA and RNA sequencing data, alongside the provision of calculating code.